CLINICAL TRIAL: NCT02649855
Title: Docetaxel and Prostvac for Metastatic Castration Sensitive Prostate Cancer
Brief Title: Docetaxel and PROSTVAC for Metastatic Castration-Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160048; 16-C-0048
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2023-07-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Prostate Neoplasms; Neoplasms, Prostatic
Keywords: PSA; Vaccine; Immunotherapy; Immune Response; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A/Sequential Docetaxel followed by PROSTVAC (Experimental): Standard androgen deprivation therapy (ADT) followed by sequential docetaxel + prostvac
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Drug: Docetaxel
- Arm B/ Combined Docetaxel with PROSTVAC (Experimental): Standard androgen deprivation therapy (ADT) followed by combined docetaxel + prostvac
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Drug: Docetaxel
- Arm C/ PROSTVAC Prior to Docetaxel (Experimental): Standard androgen deprivation therapy (ADT) followed by prostvac, then docetaxel. No ADT for less than 28 days, prostvac prior to docetaxel.
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Drug: Docetaxel

INTERVENTIONS:
Biological: PROSTVAC-V — It is a recombinant vaccinia virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules (cluster of differentiation 80 (B7.1), intercellular adhesion molecule 1 (ICAM-1), and lymphocyte function-associated antigen 3 (LFA-3). It will be given subcutaneously, 2x10(8) infectious units.
Biological: PROSTVAC-F — It is a recombinant fowlpox virus vector vaccine containing the genes for human prostate-specific antigen (PSA) and three co-stimulatory molecules (cluster of differentiation 80 (B7.1), intercellular adhesion molecule 1 (ICAM-1), and lymphocyte function-associated antigen 3 (LFA-3). It will be given subcutaneously, 1x10(9) infectious units.
Drug: Docetaxel — It is commercially available. It will be administered at 75 mg/m(2) intravenously.
  Other Names: Taxotere

SUMMARY:
Background:

Metastatic castrate-sensitive prostate cancer is cancer that has spread beyond the prostate area. It can be controlled by lowering the amount of testosterone in the body. This is called androgen deprivation therapy (ADT). The vaccine PROSTVAC might help the immune system kill cancer cells. Researchers want to add PROSTVAC and docetaxel chemotherapy to ADT. They think this may work better against prostate cancer than ADT alone.

Objective:

To test if adding PROSTVAC and docetaxel to ADT works better against prostate cancer than ADT alone.

Eligibility:

Men ages 18 years and over with metastatic castrate-sensitive prostate cancer

Design:

Participants will be screened with:

Physical exam

Medical history

Blood tests

Possible computed tomography (CT), magnetic resonance imaging (MRI), or bone scan: Participants lie in a machine. The machine takes pictures of the body.

Electrocardiogram: Soft electrodes are stuck to the skin to record heart signals.

Participants will have 2 optional tumor biopsies during the study.

Participants will join 1 of 2 groups. Both groups will get:

ADT

Docetaxel by vein

Steroids by mouth or vein before each docetaxel infusion

PROSTVAC injection

Both groups first have ADT. One to 4 months after, they have:

Group A:

Docetaxel every 3 weeks for 6 cycles

PROSTVAC 3 weeks after the last infusion

Booster injections 2 weeks later and then every 3 weeks, for 6 boosters total

Group B:

PROSTVAC

Booster 2 weeks later

Docetaxel hours later

Docetaxel and the booster every 3 weeks for 6 cycles

Participants will have a visit 4-5 weeks after the last treatment. They will then have visits every 12 weeks.

Participants will be followed for up to 15 years. This includes physical exams every year for 5 years.

DETAILED DESCRIPTION:
Background:

* A phase III trial demonstrated that combining docetaxel and androgen deprivation therapy (ADT) significantly improved survival (57.6 vs 44.0 months (hazard ration (HR)=0.56, (0.44-0.70), p <0.0001) for men with metastatic castration sensitive prostate cancer (mCSPC).
* PROSTVAC (developed by the National Cancer Institute [NCI] and licensed to Bavarian Nordic Immunotherapeutics, Mountain View, California (CA) is a therapeutic cancer vaccine for prostate cancer.
* Preclinical and clinical studies support the potential synergy in the combination of docetaxel and PROSTVAC. The potential to combine docetaxel with vaccine in mCSPC could improve upon the survival advantage that has been previously seen.

Objectives:

Primary

-To determine if PROSTVAC combined with docetaxel is able to induce greater antigen spreading (i.e. a broader immune response) with greater associated response score compared to docetaxel alone after 19 weeks.

Key Eligibility Criteria:

* Must have castrate sensitive prostate cancer (rising PSA and testosterone over 100) or is within 134 days of starting ADT (Arm A or B) or within 28 days of start ADT (Arm C)
* Histopathological confirmation of prostate cancer
* Patients must have metastatic disease
* Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria
* Patients must have adequate bone marrow, hepatic, and renal function

Design

* This is a randomized trial of ADT followed by simultaneous docetaxel 75 mg/m(2) every (q)3 weeks x 6 cycles + PROSTVAC q3 weeks x 6 cycles versus ADT followed by sequential docetaxel 75 mg/m(2) q3 weeks x 6 cycles followed by PROSTVAC q3 weeks x 6 cycles in men with newly diagnosed mCSPC.
* Patients who have not started ADT or who have been on ADT 28 days or fewer will be assigned to treatment with PROSTVAC for 4 - 6 injections followed by docetaxel 75 mg/m^2 q3 weeks x 6 cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Documented histopathological confirmation of prostate cancer-from a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory.
* Patients must have metastatic disease, defined as at least one lesion on bone scan or at least one lesion that are measurable per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. (Patients who have metastatic disease by these criteria prior to ADT, but then have changes after androgen deprivation therapy (ADT) that diminish the size of these lesions or changes on bone scan are still eligible.)
* Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria
* Patients must have adequate bone marrow, hepatic, and renal function with:

  * Absolute neutrophil count (ANC) greater than or equal to 1500/microL, without cerebrospinal fluid (CSF) support
  * Platelets greater than or equal to 100,000/microL
  * Aspartate aminotransferase (AST)/Serum glutamic-oxaloacetic transaminase (SGOT) less than or equal to 2.5 times upper limit of normal (ULN);
  * Alanine aminotransferase (ALT)/Serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 times upper limit of normal (ULN);
  * Total serum bilirubin less than or equal to 1.5 times upper limit of normal (ULN), OR in patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0)
  * Serum albumin greater than or equal to 2.8 g/dL
  * Lipase < 2.0 times the upper limit of normal and no radiologic or clinical evidence of pancreatitis
  * Creatinine less than or equal to 1.5 times institutional upper limits of normal

OR

Creatinine clearance of greater than or equal to 50 ml/min/1.73 m(2) for patients with creatinine levels above institutional normal by 24-hour urine.

* Willing to travel to the National Institutes of Health (NIH) for follow-up visits
* 18 years of age or older.
* Able to understand and sign informed consent.
* May have had up to 24 months of ADT (testosterone suppression therapy in the nonmetastatic setting) and are at least 12 months removed from treatment
* Men treated or enrolled on this protocol must also agree to use adequate contraception, prior to the study, for the duration of study participation, and 4 months after completion. Sexually active subjects and their female partners must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must also agree to use both a barrier method and a second method of birth control during the course on the study and for 4 months after the last dose of study drug(s). Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Must have started ADT for metastatic disease within 134 days (for Arm A and B) or within 28 days (for Arm C).

EXCLUSION CRITERIA:

* Immunocompromised status due to:

  * Human immunodeficiency virus (HIV) positivity.
  * Active autoimmune diseases such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Grave's disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including central nervous system (CNS), heart, lungs, kidneys, skin, and gastrointestinal (GI) tract will be allowed.
  * Other immunodeficiency diseases
* Chronic administration (defined as daily or every other day for continued use > 14 days) of corticosteroids deemed systemic by investigator within 28 days before the first planned dose of PROSTVAC. Use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed.
* Evidence of rising prostate-specific antigen (PSA) on ADT
* Serious intercurrent medical illness that, in the judgment of the investigator, would interfere with patient's ability to carry out the treatment program.
* Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (e.g. phytoestrogens and saw palmetto)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to poxviral vaccines (e.g., vaccinia vaccine)
* Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin).
* History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis
* Previous serious adverse reactions to smallpox vaccination
* Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination: (a) children less than or equal to 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczemoid skin disorders, or (d) immunocompromised individuals, such as those with human immunodeficiency virus (HIV).
* Receipt of an investigational agent within 28 days (or 60 days for an antibody-based therapy) before the first planned dose of study drugs.
* Patients who test positive for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Uncontrolled hypertension (systolic blood pressure (SBP)>170/ diastolic blood pressure (DBP)>105)
* Patients who have had prior chemotherapy for prostate cancer.
* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder).
* The subject has active brain metastases or epidural disease.
* Patients with greater than or equal to grade 2 peripheral neuropathy at baseline.
* Patients with history of splenectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0048.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
Started | 23 | 23 | 28
Completed | 19 | 19 | 25
Not Completed | 4 | 4 | 3
Not completed — Refused further treatment | 2 | 1 | 1
Not completed — Withdrew consent | 0 | 1 | 0
Not completed — Switched to alternative treatment | 0 | 1 | 1
Not completed — Principal investigator discretion | 0 | 1 | 1
Not completed — No treatment, per protocol | 1 | 0 | 0
Not completed — Initiate new treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel | Total
Number analyzed (Participants) | 23 | 23 | 28 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 12 | 13 | 17 | 42
  >=65 years | 11 | 9 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.03 (8.63) | 59.8 (14.84) | 62.81 (8.46) | 62.87 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 23 | 23 | 28 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 4 | 5
  Not Hispanic or Latino | 21 | 23 | 22 | 66
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 5 | 15
  White | 18 | 17 | 18 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 28 | 74

OUTCOME MEASURES:

1. Primary Outcome: Antigen Spreading (i.e., a Broader Immune Response) With Greater Associated Response Score Compared to Docetaxel Alone After 19 Weeks
Description: Antigen spreading as measured by antigen spread score. The antigen spreading score denotes the presence of a T-cell (cluster of differentiation(CD8)+ and/or cluster of differentiation 4(CD4+) immune response against 2 tumor associated antigens that were not targeted by PROSTVAC:Mucin 1(MUC-1) & carcinoembryonic antigen(CEA). Antigen-specific T-cell responses were determined using intracellular cytokine staining of 4 established markers (Lysosome-associated membrane proteins h-LAMP1, interferon gamma, interleukin-2& tumor necrosis factor) in both CD4+& CD8+T-cells, giving a total of 8 measures of activation per antigen. Numbers of activation markers per antigen were totaled & multiplied by 1.5 to give higher weighting to T-cell responses to antigens that were not targeted by PROSTVAC;& the scores for both MUC-1 & CEA were totaled per participant, with a possible range of 0-24 (0 is a negative result whereas 1.5-24 are positive results). The higher level of response, the better outcome.
Time Frame: After 19 Weeks
Population: 46/74 participants are evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
Number analyzed (Participants) | 16 | 12 | 18
Score on a scale | 4.31 (1.31) | 5.63 (1.63) | 4.00 (0.98)

2. Secondary Outcome: Antigen Specific T-cell Immune Composite Response Scores Between All Arms at 39 Weeks and 1 Year
Description: Response score denotes the presence of a T-cell (cluster of differentiation 8(CD8+) and/or cluster of differentiation 4(CD4+) response against 3 tumor associated antigens: prostate-specific antigen(PSA), mucin 1(MUC-1) and carcinoembryonic antigen(CEA). Antigen-specific T-cell immune responses were determined using intracellular cytokine staining of 4 established markers (Lysosome-associated membrane proteins h-LAMP1, interferon gamma, interleukin-2& tumor necrosis factor in both CD4+ & CD8+T-cells, a total of 8 measures of activation per antigen. The number of activation markers for PSA were totaled for a maximum score of 8. Numbers of activation markers for MUC-1 & CEA were totaled & multiplied by 1.5 to give higher weighting to T-cell responses to antigens that were not targeted by PROSTVAC. The scores for PSA, MUC-1 & CEA were totaled per participant, with a possible range of 0-32 (0 is a negative result whereas 1-32 are positive results). Higher level of response, better outcome.
Time Frame: 39 weeks and 1 year
Population: 46/74 participants(pts) are evaluable for this outcome measure. Analysis was not performed for Arm B at 1yr because the intent was to compare treatments when they were completed to each other in terms of immune responses. Since no further treatments were given in Arm B after the 39th week, a second analysis was not required to assess immune responses. Pts in Arms A&C may have continued treatment beyond 39 wks since they were sequential. 1yr mark was designed to capture treatments beyond wk 39.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
Number analyzed (Participants) | 16 | 12 | 18
Score on a scale
  39 Weeks | 7.03 (1.88) | 7.29 (1.83) | 6.91 (2.05)
  1 Year: number analyzed (Participants) | 16 | 0 | 18
  1 Year | 5.25 (1.48) |  | 6.44 (1.18)

3. Secondary Outcome: Number of Participants With T-cell Response to Prostate-specific Antigen (PSA)
Description: PSA-specific immune responses T-cell responses were assessed using nonparametric methods. The value denotes the number of participants with T-cell immune responses towards PSA. The higher level of response, the better outcome.
Time Frame: 39 weeks and 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
Number analyzed (Participants) | 16 | 12 | 18
Participants
  39 Weeks | 7 | 6 | 8
  1 Year: number analyzed (Participants) | 16 | 0 | 18
  1 Year | 5 |  | 13

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 70 months and 4 days for Arm A, 38 months and 28 days for Arm B, and 43 months and 29 days for Arm C.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
Number analyzed (Participants) | 23 | 23 | 28
Participants | 22 | 20 | 27

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 70 months and 4 days for Arm A, 38 months and 28 days for Arm B, and 43 months and 29 days for Arm C.
Arm/Group | Arm A/Sequential Docetaxel Followed by PROSTVAC | Arm B/ Combined Docetaxel With PROSTVAC | Arm C/ PROSTVAC Prior to Docetaxel
All-Cause Mortality (participants affected / at risk) | 11/23 | 11/23 | 6/28
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/23 | 3/28
Other Adverse Events (participants affected / at risk) | 22/23 | 20/23 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A/Sequential Docetaxel Followed by PROSTVAC (N=23) | Arm B/ Combined Docetaxel With PROSTVAC (N=23) | Arm C/ PROSTVAC Prior to Docetaxel (N=28)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A/Sequential Docetaxel Followed by PROSTVAC (N=23) | Arm B/ Combined Docetaxel With PROSTVAC (N=23) | Arm C/ PROSTVAC Prior to Docetaxel (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (3) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (11) | 6 (6) | 16 (17)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 3 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 3 (4) | 9 (9)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 4 (4) | 7 (7) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 6 (6) | 8 (8) | 15 (19)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, Eye tearing (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Eye disorders - Other, L retina abnormality (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (8) | 11 (12) | 16 (19)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 1 (1) | 5 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Broken tooth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 4 (4) | 16 (18)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 3 (3) | 5 (5) | 4 (5)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site reaction (General disorders) | 11 (14) | 14 (20) | 19 (34)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 7 (7)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 1 (1) | 6 (9)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Discolored lips- intermittent (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, sprained right ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) | 11 (12)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, numbness - right thigh (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 15 (22)
Pain in extremity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 8 (8) | 5 (5) | 3 (4)
Penile infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 11 (16)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 5 (8)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 3 (5) | 3 (7)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Abrasions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Dermatitis with rash on bilateral hands (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin-actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (5)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Watering eyes (Eye disorders) | 5 (5) | 2 (2) | 2 (2)
Weight gain (Investigations) | 2 (3) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT02649855/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02649855/ICF_001.pdf